CLINICAL TRIAL: NCT02351921
Title: Repetitive Transcranial Magnetic Stimulation in Individuals With Spinal Cord Injury: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 23423432
Record Dates: First submitted 2015-01-22; First posted 2015-01-30 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Spinal Cord Injury
Keywords: transcranial magnetic stimulation; spinal cord injury; motor cortex; somatosensory cortex
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- iTBS to primary motor cortex (Experimental): Intermittent TBS will be delivered using the 30 Hz, 600 pulse protocol targeting the primary motor cortex of the left hemisphere. The iTBS TMS coil will be placed over the motor hotspot for the representation of the flexor carpi radialis muscle.
  Interventions: Device: Transcranial magnetic stimulation
- iTBS to primary somatosensory cortex (Experimental): Intermittent TBS will be delivered using the 30 Hz, 600 pulse protocol targeting the primary motor cortex of the left hemisphere. The iTBS TMS coil will be placed over the primary somatosensory cortex located 2cm posterior to the motor hotspot for the representation of the flexor carpi radialis muscle.
  Interventions: Device: Transcranial magnetic stimulation
- Sham iTBS to primary motor cortex (Sham Comparator): Sham iTBS will be delivered using the 30 Hz, 600 pulse protocol targeting the primary motor cortex of the left hemisphere. The iTBS sham coil will be placed over the motor hotspot for the representation of the flexor carpi radialis muscle.
  Interventions: Device: Transcranial magnetic stimulation

INTERVENTIONS:
Device: Transcranial magnetic stimulation — Intermittent theta-burst stimulation is a form of repetitive Transcranial magnetic stimulation. ITBS is a non-invasive, non-painful procedure being used worldwide to study brain function and promote short-term changes (~1 hour) in neural activity in the brain. The delivery of cTBS requires ~ 40 seconds in total.
  Other Names: Repetitive TMS; intermittent theta-burst stimulation

SUMMARY:
This study will investigate how repetitive transcranial magnetic stimulation delivered as a protocol called 'continuous theta-burst stimulation (cTBS)' alters motor output and force control to a muscle in the forearm and touch perception in individuals with chronic, incomplete spinal cord injury. CTBS is a non-invasive technique that involved repetitive delivery of transcranial magnetic stimulation at a frequency of 30 Hz over the arm representation in the primary motor or sensory cortex. The purpose of this study is to determine whether cTBS is an effective intervention to increase motor output to a muscle and increase force control of that muscle and also improve the sense of touch.

DETAILED DESCRIPTION:
Experience and injury-induced neuroplasticity occur in sensory and motor pathways and cortices. Sensory and motor cortices are interconnected and collectively allow for the execution of fine, skilled hand control. Of particular interest is the role of somatosensory cortex in modulating the neural activity within primary motor cortex and ultimately influencing the control of hand movement. For somatosensory cortex to be effective in guiding hand movement it must receive an uninterrupted stream of somatosensory afferent input from skin, muscle and tendons that are active during hand movement. Damage to afferent input pathways compromise the integrity of necessary somatosensory input and contribute to impaired motor control of the hand. Following an incomplete spinal cord injury (SCI), damage to the somatosensory and motor pathways are widespread thereby compromise the integrity of afferent input that reaches somatosensory cortex [1,2]. Reducing the afferent input to somatosensory cortex leads to local changes in the concentration of GABA and promotes sensorimotor reorganization [3].

Transcranial magnetic stimulation has been used in SCI to measure residual corticospinal function [4], determine changes in the excitability of neural circuitry within the primary motor cortex [5] and induce short-lasting changes in the excitability of spinal motor neurons [6]. To date, TMS research in SCI has primarily focused on lower limb function, likely fueled by the desire to promote functional recovery of locomotion and balance control. However, one of the main determinants in promoting independent living is the ability to feed and groom oneself, relying primarily on the control of the upper limb and the dexterous use of the hand. The proposed research will investigate the ability to increase motor output to muscle of the hand and upper limb through inducing short-lasting changes within SI and investigate whether this has functional implication in force production, motor control and touch perception.

TMS may be delivered as a single, pair or a train of repetitive pulses over a particular body representation within the primary motor cortex or primary somatosensory cortex. One type of repetitive TMS is called continuous theta-burst stimulation (cTBS). The present study will deliver cTBS over the primary motor and primary somatosensory cortices in individual with chronic SCI. Measurements will be made before and following the cTBS protocol. These measures include 1) the amplitude of the motor evoked potential (MEP) that is evoked by single pulse TMS and measured in the forearm muscle, 2) force production whereby participants will be asked to perform a grip strength task where maximum force production will be measured and ability to dynamically control force production will be assessed, and 3) touch sensation whereby participants will partake in a temporal order judgment psychophysical task such that they must identify which fingertip received the tactile stimulus.

ELIGIBILITY:
Inclusion Criteria:

Individuals with chronic incomplete SCI (American spinal injury association scale B, C or D) at or below levels C4, C5, C6, C7 and T1 with injury occurring > 1 year prior will be recruited.

Exclusion Criteria:

None.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Measuring changes in motor evoked potential | Immediatately before intervention, and at 20 minutes following intervention
  The motor evoked potential is the response obtained in the forearm muscle that follows single pulse TMS. The amplitude of this measure is an indicator of the corticospinal excitability. This measure will be obtained at baseline and 20 minutes following the intervention.

SECONDARY OUTCOMES:
Measuring changes in muscle force production | Immediatately before intervention, and at 25 minutes following intervention
  Participants will be asked to squeeze a hand grip that has been fitted to a force transducer/load cell. They will be asked to maximally squeeze until a plateau is seen in the voltage output. Participants will be asked to squeeze a hand grip that has been fitted to a force transducer/load cell. They will adjust the pressure applied to the hand grip in attempt to match a random sinusoid curve that has been generated. This trial will last for 10 seconds and will be based on the maximum force generated in the previous task.

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster Unviersity, Hamilton, Ontario, Canada